CLINICAL TRIAL: NCT04758923
Title: Single-stage Versus Two-staged Management for Concomitant Gallstones and Common Bile Duct Stones
Brief Title: Management for Concomitant Gallstones and Common Bile Duct Stones.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Mahmoud Ibrahim, Resident, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Assuit university hospital..
Record Dates: First submitted 2020-09-20; First posted 2021-02-17 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Calculus Biliary
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-Stage (Active Comparator): Two-stage approach The treatment process commenced with an intial treatment phase. This will be udertaken Under General anaesthesia and entailed ERCP and endoscopic sphincterectomy
  Interventions: Procedure: Cholecystectomy
- Single stage (Active Comparator): Single stage approach Under General anaesthesia a5 trocar method will be used to access the abdominal cavity. Aconventional approach to laparoscopic cholecystectomy will be first udertaken with dissection of calot's triangle. The cystic duct will be pulled laterally to facilitate exposure of the anterior wall of the CBD, and the CBD will be opened longitudinally for a distance of approximately 1 to 1.5 cm using laparoscopic scissors. A5 mm flexible choledoscope will be used to identify the cbd stone which will be removed by flushing with sterile saline, passing a stone basket or electrohydroulic lithotripsy as neccesary to clear the CBD. A T-tube will be inserted into the CBD via the choledochotomy which will be closed by interrupted resorbable sutures before completing the cholecystectomy.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Under General anaesthesia cholecystectomy and CBD exploration

SUMMARY:
Choledocholithiasis is identified in approximately 3-10 % of patients with cholelithiasis. (1-3) While laparoscopic cholecystectomy (LC) is considered the treatment of choice in patients with gall bladder stones, there is a debate about the management of common bile duct (CBD) stones, (4) and this has led to a range of therapeutic strategies for the management of concomitant gallstones and CBD stones patients. Two-stage endoscopic management using endoscopic retrograde cholangiopancreatography (ERCP) followed by laparoscopic cholecystectomy is a common approach, although single-stage management by laparoscopic cholecystectomy with surgical exploration of the CBD is an alternative, with the single-stage approach more common in the open surgery era. Currently, it is unclear whether two-stage management is better than or at least equivalent to the single-stage surgical approach to choledocholithiasis. To address this, we undertook this study to compare these two approaches. The aim of this prospective randomized trial was to determine the best technique for the management of patients with concomitant gallstones and common bile duct stones, by comparing the success rate, complication rates, and longer-term follow-up outcomes.

DETAILED DESCRIPTION:
Single stage approach Under General anaesthesia a5 trocar method will be used to access the abdominal cavity. Aconventional approach to laparoscopic cholecystectomy will be first udertaken with dissection of calot's triangle. The cystic duct will be pulled laterally to facilitate exposure of the anterior wall of the CBDand the CBD will be opened longitudinally for adistance of approximately 1to1.5 cm using laparoscopic scissors. A5mm flexible choledoscope will be used to identify the CBD stone(s) which will be removed by flushing sterile saline, passingastone basket, or electrohydraulic lithotrpsy as necessary to clear the CBD. A T-tube will be inserted into the CBD via the choledochotomy which will be closed by interrupted resorbable sutures, before completing the cholecystectomy. Cholangiography throuh T-tube be performed 14 14 days later and the T-tube will be removed immediately after Cholangiography if no residual CBD stones is identified. If residual stones are found then will be removed through the T-tube track using A choledoscope Two-stage approach The treatment process commenced with intial endoscopic treatment phase. This will be udertaken Under General anaesthesia and entailed ERCP and endoscopic sphincterectomy. The CBD stones will be removed using a basket or ballon, with lithotrpsy added if necessary. An endoscopic nasobiliary drainge will be inserted and kept in place until after laparoscopic cholecystectomy which perfermed 2 to 5 days later depending on the patients 's condition.. Surgery will be delsyed if urine amylase is elevated or significant abdominal pain is present. 2 to 5 days after the operation, Cholangiography will be performed via endoscopic nasobiliary drainge tube. And the endoscopic nasobiliary drainge tube wii be removed if no residual CBD stones are seen.

ELIGIBILITY:
Inclusion Criteria:

Age 16 to 70 years; Clinical presentation with biliary colic with or without jaundice; Serum elevation of at least one of the following enzymes: aspartate aminotransferase, alanine aminotransferase, glutamyl transpeptidase, alkaline phosphatase, and total bilirubin; Radiological findings suggestive of gallstones and concomitant common bile duct stones, with abdominal ultrasound showing possible CBD stones or a dilated CBD >8 mm in diameter.

only patients with MRCP evidence of a CBD stone(s) were eligible after meeting all the previous criteria.

Exclusion Criteria:

active acute pancreatitis, pregnancy, septic shock, intrahepatic gallstones, malignant pancreatic or biliary tumors, prior sphincterotomy, unfit for anesthesia and surgery, contraindications to MRCP and ERCP, liver cirrhosis, previous history of abdominal surgery (e.g., gastrectomy), and inability to give informed consent.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical successful rates | 2 weeks
  The prospective clinical trial aims to determine the best technigue for the management of the patient with concomitant GB and CBD stones by comparing success rate and complication rates

IPD SHARING:
Plan to Share IPD: No